CLINICAL TRIAL: NCT02896374
Title: Normal and Abnormal Event Related Potentials During Attribution of Intentions to Others and Resolution of Emotional Conflicts in Schizophrenia
Brief Title: Normal and Abnormal ERP During ToM and Emotional Conflicts in Schizophrenia
Acronym: SERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Eric BRUNET, Investigator coordinator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P11/16_SERC
Record Dates: First submitted 2016-08-19; First posted 2016-09-12 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Treated or hospitalized patients for schizophrenia.
  Interventions: Behavioral: Theory of mind without visual cues
- Control (Experimental): No schizophrenic participants, comparable to schizophrenia patients in age, gender, education level and socio premorbid verbal IQ.
  Interventions: Behavioral: Theory of mind without visual cues

INTERVENTIONS:
Behavioral: Theory of mind without visual cues — Theory of mind stimulation without visual reinforcement while performing EEG recordings
Behavioral: Theory of mind without visual cues — Theory of mind stimulation with visual reinforcement while performing EEG recordings

SUMMARY:
Case-control comparison of clinical population, interventional and single-center research.

DETAILED DESCRIPTION:
The main objective of this study is to define and characterize electrophysiological markers of the existing social cognition disorders in schizophrenia. Two groups of subjects are recorded : schizophrenic patients and healthy controls. Visual reinforcement effect during theory of mind judgment is tested.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent French mother tongue Schizophrenia diagnosis according to DSM-IV-R for the patient group

Exclusion Criteria:

Coma history, epilepsy, head trauma with loss knowledge greater 10 min ECT older than 1 month DSM-4 R criteria of toxic addiction in the last 6 months Deafness or blindness Scalp pathology Intracranial implanted device

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Event related electric amplitudes | Day 0
  Scalp EEG recordings (microvolts) with respect to average or vertex references

CONTACTS AND LOCATIONS:
Overall Officials: Eric Brunet, MD PhD, Principal Investigator — Versailles Hospital
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: Undecided